CLINICAL TRIAL: NCT06049771
Title: The Population Pharmacokinetics Study of Tigecycline and Pharmacokinetics- Pharmacodynamics Index in Patients With Carbapenem Resistant Enterobacteriaceae Bloodstream Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Silpakorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMK0009
Record Dates: First submitted 2023-07-31; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Carbapenem-resistant Enterobacteriaceae
Keywords: Tigecycline; Population pharmacokinetics; pharmacokinetics-pharmacodynamics index; bloodstream infection; CRE; Carbapenem-resistant Enterobacteriaceae
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Patients who were infected caused by CRE bloodstream infection and were treated with tigecycline. Blood samples were collected.
  Interventions: Other: Collect blood sample

INTERVENTIONS:
Other: Collect blood sample — Collect blood samples at different time points: after tigecycline administration 1 h, 2-4 h, 4-6 h, 6-11.5 h and 30 minutes before next dose

SUMMARY:
Carbapenem-resistant Enterobacteriaceae (CRE) are an urgent global public health problem. Patients who were infected caused by CRE bloodstream infection were high mortality up to 40%. The National Antimicrobial Resistance Surveillance Center, Thailand (NARST) reported CRE increased from 1.1% to 17.9%. For carbapenemase producing CRE in Thailand was reported blaNDM 47.33%, blaOXA-48 43.33% and blaNDM+blaOXA-48 6.67%.

Tigecycline (TGC) was a glycylcyclines antibiotics. High dose tigecycline (HD-TGC) loading dose 200 mg then TGC 100 mg q 12 h via intravenous improve clinical cure in critically ill patients and reduce mortality in carbapenem resistance Klebsiella pneumoniae bloodstream infection compared with standard dose therapy. TGC has susceptibility to CR-KP 79.6% and has an activity to blaNDM, blaKPC and blaOXA-48 carbapenemase producing CRE. However, TGC has clearance (CL) 0.2-0.3 L/h/kg, and high volume of distribution (vd) 2.8-13 L/kg resulted in low levels of TGC in plasma. Moreover, the pharmacokinetics of TGC in critically ill was limited and inconsistent with the previous study. Now pharmacokinetics-pharmacodynamics index (PK/PD index) of TGC for CRE bloodstream infection was not reported. This study aims to study the population pharmacokinetic and PK-PD index of TGC in patients who were CRE bloodstream infection to increase the success rate of treatment.

DETAILED DESCRIPTION:
Carbapenem-resistant Enterobacteriaceae (CRE) are an urgent global public health problem. Patients who were infected caused by CRE bloodstream infection were high mortality up to 40%. The National Antimicrobial Resistance Surveillance Center, Thailand (NARST) reported the carbapenem resistance Klebsiella pneumoniae (CR-KP) prevalence increased from 1.1% in 2000 to 17.9% in 2021 and the carbapenem resistance Escherichia coli was increased from 0.6% in 2000 to 5% in 2021. For carbapenemase producing CRE in Thailand was reported blaNDM 47.33%, blaOXA-48 43.33%, and blaNDM+blaOXA-48 6.67%. Ceftazidime-avibactam was first-line of treatment for CRE bloodstream infection recommended by Infectious Disease Society of America 2023 guidance on the treatment of antimicrobial resistant gram-negative infections but ceftazidime-avibactam was limited activity to blaNDM carbapenemase producing CRE.

Tigecycline (TGC) was a glycylcyclines antibiotics. TGC was approved for U.S.FDA for complicated intra-abdominal infection, complicated skin and skin structure infection and community acquired pneumonia with loading dose TGC 100 mg then TGC 50 mg q 12 h via intravenous. High dose tigecycline (HD-TGC) loading dose 200 mg then TGC 100 mg q 12 h improve clinical cure in critically ill patients and reduce mortality in CR-KP bloodstream infection compared with standard dose therapy. TGC has susceptibility to CR-KP 79.6% and has an activity to blaNDM, blaKPC and blaOXA-48 carbapenemase producing CRE. However, TGC has clearance (CL) 0.2-0.3 L/h/kg, and high volume of distribution (vd) 2.8-13 L/kg resulted in low levels of TGC in plasma. Moreover, the pharmacokinetics of TGC in critically ill was limited and inconsistent with the previous study. Now pharmacokinetics-pharmacodynamics index (PK/PD index) of TGC for CRE bloodstream infection was not reported. This study aims to study the population pharmacokinetic and PK-PD index of TGC in patients who were CRE bloodstream infection to increase the success rate of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years and older who were admitted at Phramongkutklao Hospital
2. Patients who were diagnosed bloodstream infection with CRE and who were sepsis or septic shock
3. Patients who received tigecycline loading dose 200 mg infusion for 1 hour and following maintenance dose 100 mg every 12 h infusion for 1 hour at least 48 hours and grant for blood collection

Exclusion Criteria:

1. Pregnancy or Breastfeeding
2. Patients who cannot tolerant to the toxicity of tigecycline for example hypersensitivity to tigecycline or any component of the formulation
3. Patients who were infected with more than one isolated in blood culture at the same time

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-09-17 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
rate constant for tigecycline distribution from the central to the peripheral compartment | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline
rate constant for tigecycline distribution from the peripheral to central the compartment | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline
elimination rate constant | up to 6 months
  Population pharmacokinetic parameter of tigecycline
intercompartmental clearance | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline
total clearance | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline
volume of central compartment | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline
volume distribution of peripheral compartment | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline
steady state volume distribution | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline
Area under the plasma concentration versus time curve (AUC) | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline
Peak Plasma Concentration (Cmax) | up to 6 months
  Population pharmacokinetic parameter outcome of tigecycline

SECONDARY OUTCOMES:
PK/PD index for CRE bloodstream infection | up to 6 months
  pharmacokinetics-pharmacodynamics parameter of tigecycline for CRE bloodstream infection
Rate of mortality | 7,14 and 28 days
  Alive or death
Number of Participants with the clinical outcome | 14 days
  Clinical cure or clinical failure Clinical cure was defined as the resolution or improvement of all signs and symptoms present at study entry Clinical failure was defined as any one or more following circumstances: persistent or worsened signs and symptoms, a new clinical findings consistent with the progression of infection.
Number of Participants with the microbiological outcome | 7 days
  Eradicated or persistent evaluated by culture of bloodstream
Genotype classification of carbapenemase producing CRE | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sirapat Somsirikarnjanakoon, PharmD., Study Chair — Faculty of Pharmacy, Silpakorn University; Wichai Santimaleeworagun, PhD., Study Director — Faculty of Pharmacy, Silpakorn University; Worapong Nasomsong, MD., Study Director — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramongkutklao Hospital, Ratchathewi, Bangkok, Thailand